CLINICAL TRIAL: NCT06862661
Title: Enhancing Breastfeeding Self-Efficacy in Filipino Mothers: Assessing the Impact of the LactApp m-Health Tool
Acronym: A Mixed-Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angeles University Foundation (Other)
Responsible Party: Principal Investigator, Rudena A. Madayag, Assistant Professor, Angeles University Foundation
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2024-CON-Faculty-004; 2024-CON-Faculty-004 (Other: Angeles University Foundation Ethics Review Committee)
Record Dates: First submitted 2025-02-20; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Breastfeeding Education
Keywords: Breastfeeding practices; Breastfeeding self-efficacy; Lactation Support; Maternal Health; Mobile Health Applications

STUDY DESIGN:
Intervention Model Description: The intervention involves introducing the LactApp tool to mothers to enhance breastfeeding self-efficacy. Researchers assist participants in downloading and navigating the app, which offers features like daily breastfeeding tips, tracking tools, and expert support. Mothers are encouraged to use the app regularly, with weekly follow-ups to monitor engagement and provide additional support, aiming to improve their breastfeeding experience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impact of LactApp on Breastfeeding Self-Efficacy in Filipino Mothers (Experimental): This study focuses on evaluating the impact of the LactApp mobile application on the breastfeeding self-efficacy of Filipino mothers. Participants will complete a pre-test survey using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) to establish baseline confidence levels in breastfeeding. They then used the LactApp tool for 3 months, which provided personalized advice, tracking tools, and educational content. After the intervention, the same survey will be administered as a post-test to measure changes in self-efficacy.
  Interventions: Other: Daily Tips and Advice on the use of LactApp m-health tool throughout the breastfeeding journey.

INTERVENTIONS:
Other: Daily Tips and Advice on the use of LactApp m-health tool throughout the breastfeeding journey. — A tool to track breastfeeding frequency, duration, and baby's weight and offers access to a community forum for peer support along with direct consultations with lactation experts.
  Other Names: Tracking Tool.

SUMMARY:
This study aimed to evaluate the effectiveness of LactApp in improving breastfeeding self-efficacy among Filipino mothers.

DETAILED DESCRIPTION:
Breastfeeding is crucial for maternal and child health, but Filipino mothers face significant challenges, worsened by the COVID-19 pandemic, which has limited access to traditional breastfeeding support. This study proposes evaluating the LactApp mobile application as a tool to enhance breastfeeding self-efficacy among Filipino mothers and improve nursing education.

The study's objectives include assessing LactApp's effectiveness in boosting mothers' confidence in breastfeeding and identifying gaps in nursing students' breastfeeding education. A mixed-methods approach will be used, combining quantitative assessments (via the Breastfeeding Self-Efficacy Scale-Short Form) and qualitative focus group discussions with mothers and nursing students. The study will also analyze user engagement and common breastfeeding queries to tailor educational content.

Expected outcomes include empowering nursing students with better breastfeeding knowledge, improving maternal support, and integrating digital tools like LactApp into nursing curricula. Ultimately, the study aims to enhance breastfeeding outcomes for Filipino mothers and contribute to improved maternal and child health in the community.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 16-45, including those who are pregnant or have recently given birth (within the last 12 months).
* Females who are currently seeking breastfeeding support and are open to using the LactApp tool.
* Females who are willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Females who are not intending to breastfeed.
* Females with significant health issues that may impair their ability to use the LactApp tool or participate in the study.
* Females who are not fluent in the language in which the LactApp tool is provided, making it difficult for them to engage with the content.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Filipino mothers who were either pregnant or had children under the age of one, was specifically chosen because these groups are most directly impacted by the challenges of breastfeeding and maternal health, and they are the ideal demographic for studying the effectiveness of breastfeeding interventions such as the LactApp tool.
Enrollment: 280 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in breastfeeding self-efficacy | From enrollment to the end of the intervention at 3 months
  The primary outcome of this study is the enhancement of breastfeeding self-efficacy among Filipino mothers following the use of the LactApp mobile Health tool. This outcome is measured using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), a validated tool designed to assess a mother's confidence in her ability to breastfeed. The BSES-SF consists of 14 items, each scored on a 5-point Likert scale ranging from 1 ("Not at all confident") to 5 ("Always confident"). The total score ranges from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy. This scale is widely used in maternal health research to evaluate interventions aimed at improving breastfeeding outcomes.

SECONDARY OUTCOMES:
Maternal Confidence in Breastfeeding | Four weeks after intervention to the end of 3 months.
  Assesses mothers' self-reported confidence in initiating and sustaining breastfeeding. Data will be collected through semi-structured interviews.
Decision-Making in Breastfeeding Practices | Four weeks after intervention to the end of 3 months.
  Evaluates the factors influencing mothers' feeding decisions, including the role of informational support provided by LactApp. Data will be collected through semi-structured interviews.
Sense of Empowerment | Four weeks after intervention to the end of 3 months.
  Assess the extent to which breastfeeding contributes to mothers' feelings of autonomy and overall empowerment in managing their infant's feeding. Data will be collected through semi-structured interviews.
Identification of Barriers | Four weeks after intervention to the end of 3 months.
  Identifies potential barriers to effective use of the LactApp, including issues related to digital literacy and accessibility, which may impact breastfeeding self-efficacy. Data will be collected through semi-structured interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Angeles University Foundation, Mac Arthur Highway, Angeles City, Pampanga, Philippines

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: Access to Individual Participant Data (IPD) and supporting information from the study will be granted to researchers, healthcare professionals, and policymakers with a legitimate interest in maternal healthcare. Interested individuals must demonstrate a clear research purpose, such as conducting secondary analyses or developing new interventions. Authorized users will access anonymized IPD, including demographic information and breastfeeding self-efficacy scores, while ensuring participant privacy. Supporting documentation will consist of the study protocol and data collection tools. Access will be managed through a data-sharing agreement to ensure ethical use. Interested parties must submit a formal request outlining their objectives, which will be reviewed by a data-sharing committee. Once approved, users can access the data via a secure online platform, ensuring responsible utilization that advances research and improves maternal healthcare outcomes.